CLINICAL TRIAL: NCT03561220
Title: A Prospective Comparative Study of Outcomes With Proton and Photon Radiation in Prostate Cancer
Acronym: COMPPARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMPPARE; PCORI-6312 (Other Grant/Funding Number: PCORI); IRB201801001 (Other: University of Florida); OCR17881 (Other: University of Florida)
Record Dates: First submitted 2018-05-15; First posted 2018-06-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Proton Radiation; Photon Radiation; Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IMRT (Photon) (Active Comparator): As this trial is pragmatic, all treatment will be standard of care.
  Interventions: Radiation: Standard of Care IMRT (Photon)
- Proton Therapy Standard of Care (Active Comparator): As this trial is pragmatic, all treatment will be standard of care.
  Interventions: Radiation: Standard of Care Proton Therapy
- Standard Proton Therapy (Experimental): 78.0 Gy (RBE) in 39 fractions. This is Arm 1 of the embedded randomized trial.
  Interventions: Radiation: Proton Arm 1: Standard Proton Therapy
- Hypofractionated Proton therapy (Experimental): 60.0 Gy (RBE) in 20 fractions This is Arm 2 of the embedded randomized trial.
  Interventions: Radiation: Proton Arm 2: Hypofractionated Proton Therapy

INTERVENTIONS:
Radiation: Standard of Care IMRT (Photon) — As this trial is pragmatic, all treatment will be standard of care.
  Arms: IMRT (Photon)
Radiation: Standard of Care Proton Therapy — As this trial is pragmatic, all treatment will be standard of care.
  Arms: Proton Therapy Standard of Care
Radiation: Proton Arm 1: Standard Proton Therapy — 78.0 Gy (RBE) in 39 fractions
  Arms: Standard Proton Therapy
Radiation: Proton Arm 2: Hypofractionated Proton Therapy — 60.0 Gy (RBE) in 20 fractions
  Arms: Hypofractionated Proton therapy

SUMMARY:
This study is a large, prospective, pragmatic, controlled comparison of patient-centric outcomes [quality of life (QOL), toxicity, and disease control] between parallel cohorts of men with prostate cancer treated simultaneously at proton therapy facilities and at geographically similar conventional (photon-based) radiation facilities using intensity-modulated radiation therapy (IMRT) techniques.

DETAILED DESCRIPTION:
This study is a large, prospective, pragmatic, controlled comparison of patient-centric outcomes [quality of life (QOL), toxicity, and disease control] between parallel cohorts of men with prostate cancer treated simultaneously at proton therapy facilities and at geographically similar conventional (photon-based) radiation facilities using intensity-modulated radiation therapy (IMRT) techniques. This study includes a pre-specified randomized comparison of standard fractionation and moderate hypofractionation dose schemes within the proton therapy cohort. In addition, subgroup analyses will include a comparison of outcomes by race (Black vs. White), comorbidity score (0 vs. 1+), age (<65 vs. ≥65), fractionation schedule (standard, moderate, ultra-hypofractionation), and prostate cancer aggressiveness (very low and low, intermediate, and high risk) for all objectives.

All interventions will be standard of care (SOC) radiation strategies using either IMRT or proton therapy. All patient-reported QOL, patient-scored and patient-reported toxicity, and disease control assessments will be SOC. Participants will also complete pretreatment surveys regarding demographic data, personal treatment goals, factors affecting treatment decision-making, and sources of information used in treatment selection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the prostate.
* 30-85 years of age at the time of consent with a life expectancy estimation (LEE) of ≥ 8 years.
* Localized prostate cancer, as confirmed by staging with PSA, biopsy, Gleason score, DRE with or without mpMRI, and clinical stage.
* Very low-risk, low-risk, intermediate-risk, or high-risk disease based on NCCN Prostate Cancer Risk Group Guidelines and Joint AUA/ASTRO/SUO Guidelines.
* If patient has high-risk disease, nuclear medicine bone imaging must be performed to document the absence of overt metastatic disease in bones.
* ECOG/Zubrod Performance Status 0 - 2.
* Candidate for definitive prostate radiotherapy (either IMRT or proton).
* If patient is to be treated with IMRT, all treatment must be planned with IMRT; if patient is to be treated with protons, all treatment must be planned with protons (including pelvic nodes if treated).

Exclusion Criteria:

* Findings of metastatic disease (nodal or distant, N1 or M1).
* Very high-risk prostate cancer based on NCCN Prostate Cancer Risk Group Guidelines and Joint AUA/ASTRO/SUO Guidelines.
* Prior procedures for treatment of prostate cancer, such as radical or robotic prostatectomy, high-intensity focused ultrasound, cryosurgery, or focal prostatectomy [note that procedures used for benign prostatic hyperplasia symptoms, such as transurethral resection of the prostate (TURP) and GreenLight Laser Therapy, are acceptable].
* Previous prostate cancer treatment with the exception of ADT according to NCCN guidelines.
* History of invasive rectal malignancy or other malignancy in the true pelvis (e.g. bladder, rectum, or reproductive organs), regardless of disease-free interval.
* Active inflammatory bowel disease (i.e., patients requiring medical interventions or who are symptomatic).
* Prior pelvic RT for any reason.
* Documented lack of psychological ability or general health permitting completion of the study requirements and required follow-up.
* Documented diminished capacity to understand the risks and benefits of participation in research and to autonomously provide informed consent.

In addition, because the embedded randomized controlled trial compares fractionation schemes, patients who are receiving pelvic node irradiation may not be enrolled on the randomized controlled trial.

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2018-07-05 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Bowel urgency and bowel frequency Expanded Prostate Cancer Index Composite (EPIC) item scores | 2-years after the end of radiation therapy
  EPIC assesses the disease-specific aspects of prostate cancer and its therapies and comprises four summary domains (Urinary, Bowel, Sexual and Hormonal). Factor analysis supports dividing the Urinary Domain Summary Score into two distinct Incontinence and Irritative/Obstructive subscales. In addition, each Domain Summary Score has measurable Function Subscale and Bother Subscale components. Response options for each EPIC item form a Likert scale, and multi-item scale scores are components. Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL

SECONDARY OUTCOMES:
Grade 2 or higher toxicity for each adverse event assessed by CTCAE | 2-years after the end of radiation therapy
  The NCI Common Terminology Criteria for Adverse Events v5.0 is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.
Grade 2 or higher toxicity for each adverse event assessed by PRO-CTCAE. | 2-years after the end of radiation therapy
  PRO-CTCAE responses are scored from 0 to 4, and there are as yet no standardized scoring rules for how to combine attributes into a single score or how best to analyse PRO-CTCAE data longitudinally. PRO-CTCAE scores for each attribute (frequency, severity and/or interference) should be presented descriptively (e.g. summary statistics or graphical presentations). CTCAE grades for the corresponding time period should be presented in conjunction with PRO-CTCAE scores.
Freedom from biochemical progression using PSA results. | 3-years after the end of radiation therapy
  Biochemical failure is defined as a sustained rise in PSA of 2 ng/mL or more above the nadir (the lowest PSA level after radiotherapy).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy P. Mendenhall, MD, Principal Investigator — University of Florida
Locations (53):
- United States (53):
  - University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - Proton Therapy Treatment Center - Loma Linda University, Loma Linda, California
  - Sutter Health, Roseville, California
  - California Protons Cancer Therapy Center, San Diego, California
  - Department of Radiation Oncology Davis Cancer Pavilion, Gainesville, Florida
  - University of Florida Proton Therapy Institute, Jacksonville, Florida
  - Ackerman Cancer Center, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health UF Health Center, Orlando, Florida
  - Winship Cancer Institute - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Northwestern Medicine Proton Center, Warrenville, Illinois
  - University of Kansas Medical Center, Lawrence, Kansas
  - University of Louisville, Louisville, Kentucky
  - Willis-Knighton Medical Center PTC, Shreveport, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland, College Park, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Health System, Mankato, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - S Lee Kling Proton Therapy Center - Washington University Medical Center, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Covenant Health, Somerset, New Jersey
  - New York Proton Center, New York, New York
  - Weill Cornell, New York, New York
  - The Duke University Health System, Durham, North Carolina
  - UNC- Rex Hospital, Raleigh, North Carolina
  - University of Cincinnati Medical PTC, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals- Seidman Cancer Center, Cleveland, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania--Penn Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Provision CARES Proton Therapy Center Knoxville, Knoxville, Tennessee
  - Texas Oncology, Austin, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Center for Proton Therapy, Irving, Texas
  - Texas Oncology - Longview, Longview, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology - Plano West, Plano, Texas
  - Texas Oncology - Waco, Waco, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Hampton University Proton Therapy Institute, Hampton, Virginia
  - Seattle Care Alliance/University of Washington, Seattle, Washington
  - Mayo Clinic Health System, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, Sparta, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NCCN Clinical Practical Guidelines in Oncology: Prostate Cancer. Version 2. 2018.
- [Background] AJCC Cancer Staging Manual. 8th ed. Cham, Switzerland: Springer International Publishing; 2017.
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] U.S. Preventive Services Task Force. Draft Recommendation Statement: Prostate Cancer: Screening. April 2017; https://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatementDraft/prostate-cancer-screening1. Accessed May 8, 2017.
- [Background] Chen RC, Clark JA, Talcott JA. Individualizing quality-of-life outcomes reporting: how localized prostate cancer treatments affect patients with different levels of baseline urinary, bowel, and sexual function. J Clin Oncol. 2009 Aug 20;27(24):3916-22. doi: 10.1200/JCO.2008.18.6486. Epub 2009 Jul 20. PMID 19620493
- [Background] Sanda MG, Dunn RL, Michalski J, Sandler HM, Northouse L, Hembroff L, Lin X, Greenfield TK, Litwin MS, Saigal CS, Mahadevan A, Klein E, Kibel A, Pisters LL, Kuban D, Kaplan I, Wood D, Ciezki J, Shah N, Wei JT. Quality of life and satisfaction with outcome among prostate-cancer survivors. N Engl J Med. 2008 Mar 20;358(12):1250-61. doi: 10.1056/NEJMoa074311. PMID 18354103
- [Background] Stokes ME, Ishak J, Proskorovsky I, Black LK, Huang Y. Lifetime economic burden of prostate cancer. BMC Health Serv Res. 2011 Dec 28;11:349. doi: 10.1186/1472-6963-11-349. PMID 22204308
- [Background] Riley GF, Potosky AL, Lubitz JD, Kessler LG. Medicare payments from diagnosis to death for elderly cancer patients by stage at diagnosis. Med Care. 1995 Aug;33(8):828-41. doi: 10.1097/00005650-199508000-00007. PMID 7637404
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Gray PJ, Lin CC, Cooperberg MR, Jemal A, Efstathiou JA. Temporal Trends and the Impact of Race, Insurance, and Socioeconomic Status in the Management of Localized Prostate Cancer. Eur Urol. 2017 May;71(5):729-737. doi: 10.1016/j.eururo.2016.08.047. Epub 2016 Sep 3. PMID 27597241
- [Background] Miller KD, Siegel RL, Lin CC, Mariotto AB, Kramer JL, Rowland JH, Stein KD, Alteri R, Jemal A. Cancer treatment and survivorship statistics, 2016. CA Cancer J Clin. 2016 Jul;66(4):271-89. doi: 10.3322/caac.21349. Epub 2016 Jun 2. PMID 27253694
- [Background] Chamie K, Williams SB, Hu JC. Population-Based Assessment of Determining Treatments for Prostate Cancer. JAMA Oncol. 2015 Apr;1(1):60-7. doi: 10.1001/jamaoncol.2014.192. PMID 26182305
- [Background] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Background] Zietman A. Proton beam and prostate cancer: An evolving debate. Rep Pract Oncol Radiother. 2013 Jul 3;18(6):338-42. doi: 10.1016/j.rpor.2013.06.001. PMID 24416575
- [Background] Wisenbaugh ES, Andrews PE, Ferrigni RG, Schild SE, Keole SR, Wong WW, Vora SA. Proton beam therapy for localized prostate cancer 101: basics, controversies, and facts. Rev Urol. 2014;16(2):67-75. PMID 25009446
- [Background] Vargas C, Fryer A, Mahajan C, Indelicato D, Horne D, Chellini A, McKenzie C, Lawlor P, Henderson R, Li Z, Lin L, Olivier K, Keole S. Dose-volume comparison of proton therapy and intensity-modulated radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):744-51. doi: 10.1016/j.ijrobp.2007.07.2335. Epub 2007 Sep 27. PMID 17904306
- [Background] Trofimov A, Nguyen PL, Coen JJ, Doppke KP, Schneider RJ, Adams JA, Bortfeld TR, Zietman AL, Delaney TF, Shipley WU. Radiotherapy treatment of early-stage prostate cancer with IMRT and protons: a treatment planning comparison. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):444-53. doi: 10.1016/j.ijrobp.2007.03.018. Epub 2007 May 21. PMID 17513063
- [Background] Friedland W, Schmitt E, Kundrat P, Dingfelder M, Baiocco G, Barbieri S, Ottolenghi A. Comprehensive track-structure based evaluation of DNA damage by light ions from radiotherapy-relevant energies down to stopping. Sci Rep. 2017 Mar 27;7:45161. doi: 10.1038/srep45161. PMID 28345622
- [Background] Winter M, Dokic I, Schlegel J, Warnken U, Debus J, Abdollahi A, Schnolzer M. Deciphering the Acute Cellular Phosphoproteome Response to Irradiation with X-rays, Protons and Carbon Ions. Mol Cell Proteomics. 2017 May;16(5):855-872. doi: 10.1074/mcp.M116.066597. Epub 2017 Mar 16. PMID 28302921
- [Background] Grosse N, Fontana AO, Hug EB, Lomax A, Coray A, Augsburger M, Paganetti H, Sartori AA, Pruschy M. Deficiency in homologous recombination renders Mammalian cells more sensitive to proton versus photon irradiation. Int J Radiat Oncol Biol Phys. 2014 Jan 1;88(1):175-81. doi: 10.1016/j.ijrobp.2013.09.041. Epub 2013 Nov 13. PMID 24239385
- [Background] Tommasino F, Durante M. Proton radiobiology. Cancers (Basel). 2015 Feb 12;7(1):353-81. doi: 10.3390/cancers7010353. PMID 25686476
- [Background] Bryant C, Smith TL, Henderson RH, Hoppe BS, Mendenhall WM, Nichols RC, Morris CG, Williams CR, Su Z, Li Z, Lee D, Mendenhall NP. Five-Year Biochemical Results, Toxicity, and Patient-Reported Quality of Life After Delivery of Dose-Escalated Image Guided Proton Therapy for Prostate Cancer. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):422-434. doi: 10.1016/j.ijrobp.2016.02.038. Epub 2016 Feb 16. PMID 27084658
- [Background] Mendenhall NP, Hoppe BS, Nichols RC, Mendenhall WM, Morris CG, Li Z, Su Z, Williams CR, Costa J, Henderson RH. Five-year outcomes from 3 prospective trials of image-guided proton therapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2014 Mar 1;88(3):596-602. doi: 10.1016/j.ijrobp.2013.11.007. PMID 24521677
- [Background] Waddle MR, Sio TT, Van Houten HK, Foote RL, Keole SR, Schild SE, Laack N, Daniels TB, Crown W, Shah ND, Miller RC. Photon and Proton Radiation Therapy Utilization in a Population of More Than 100 Million Commercially Insured Patients. Int J Radiat Oncol Biol Phys. 2017 Dec 1;99(5):1078-1082. doi: 10.1016/j.ijrobp.2017.07.042. Epub 2017 Aug 2. PMID 28939229
- [Background] Resnick MJ, Koyama T, Fan KH, Albertsen PC, Goodman M, Hamilton AS, Hoffman RM, Potosky AL, Stanford JL, Stroup AM, Van Horn RL, Penson DF. Long-term functional outcomes after treatment for localized prostate cancer. N Engl J Med. 2013 Jan 31;368(5):436-45. doi: 10.1056/NEJMoa1209978. PMID 23363497
- [Derived] Liu Y, Patel SA, Jani AB, Gillespie TW, Patel PR, Godette KD, Hershatter BW, Shelton JW, McDonald MW. Overall Survival After Treatment of Localized Prostate Cancer With Proton Beam Therapy, External-Beam Photon Therapy, or Brachytherapy. Clin Genitourin Cancer. 2021 Jun;19(3):255-266.e7. doi: 10.1016/j.clgc.2020.08.009. Epub 2020 Aug 28. PMID 32972877